CLINICAL TRIAL: NCT03321318
Title: AK-R215 Pharmacokinetic Study Pharmacokinetic Characteristics of AK-R215 in Comparison to Each Component Coadministered in Healthy Adult Male or Menopausal Female Valunteers.
Brief Title: AK-R215 Pharmacokinetic Study Phase I
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AK-CTR-215-I-02
Record Dates: First submitted 2017-07-19; First posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Healthy
MeSH Terms: interventions — bazedoxifene; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group (Experimental): AK-R215, test drug
  Interventions: Drug: AK-R215; Drug: Bazedoxifene 20 mg; Drug: Cholecalciferol 800IU
- B group (Active Comparator): reference drug, Bazedoxifene 20mg, Cholecalciferol 800IU
  Interventions: Drug: AK-R215; Drug: Bazedoxifene 20 mg; Drug: Cholecalciferol 800IU

INTERVENTIONS:
Drug: AK-R215 — Investigational product is prescribed to all ofrandomized subjects
Drug: Bazedoxifene 20 mg — Investigational product is prescribed to all of randomized subjects
Drug: Cholecalciferol 800IU — Investigational product is prescribed to all of randomized subjects

SUMMARY:
An open label, randomized, 2-sequence, 2-period, single-dose cross-over study to evaluate the pharmacokinetics characteristics of AK-R215

DETAILED DESCRIPTION:
An open label, randomized, 2-sequence, 2-period, single-dose cross-over study to evaluate the safety and pharmacokinetics characteristics after administration of fixed dose combination or loose combination of AK-R215 in healthy adult male or menopausal female volunteers

ELIGIBILITY:
Inclusion Criteria:

* BW is above 50kg and BMI is between 18.5 and 30.0
* Subject who agreed and signed on informed consent form prior to the study participation

Exclusion Criteria:

* Presence or history of clinically significant disease
* Treatment history of any drug which might affect IP within 10days
* History of other study drugs within 12weeks

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-07-13 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2018-01-12 (Estimated)

PRIMARY OUTCOMES:
AUC0-t | 0, 0.25, 0.5, 1, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 60, 72, 96, 120h
Cmax | 0, 0.25, 0.5, 1, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 60, 72, 96, 120h

SECONDARY OUTCOMES:
Tmax | 0, 0.25, 0.5, 1, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 60, 72, 96, 120h
AUCinf, | 0, 0.25, 0.5, 1, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 60, 72, 96, 120h
T1/2 | 0, 0.25, 0.5, 1, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 60, 72, 96, 120h

CONTACTS AND LOCATIONS:
Locations (1):
- Dong-A University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided